CLINICAL TRIAL: NCT04795414
Title: Safety and Immunogenicity of an Inactivated Vaccine Against COVID-19 in Medical Workers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RJHKY2021-12
Record Dates: First submitted 2021-03-11; First posted 2021-03-12 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV-2 Infection; Covid19
Keywords: SARS-CoV-2; Covid19; Inactivated vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, including plasma, serum and blood cell
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccination Group: Participants vaccinated with inactivated SARS-CoV-2 vaccine are studied for safety and antibody response.
  Interventions: Biological: SARS-CoV-2 Vaccine(Vero Cell), Inactivated

INTERVENTIONS:
Biological: SARS-CoV-2 Vaccine(Vero Cell), Inactivated — The subjects of Vaccination Group will receive two doses, 21 days apart of inactivated SARS-CoV-2 vaccine (4 μg of BBIBP-CorV)

SUMMARY:
With the unprecedented morbidity of the COVID-19 pandemic, the vaccine effectiveness needs to be assessed across diverse populations. The purpose of this study is to evaluate the safety and immunogenicity of an inactivated SARS-CoV-2 vaccine in medical workers.

DETAILED DESCRIPTION:
1370 participants who were negative for serum-specific antibodies against SARS-CoV-2 at the time of screening were enrolled and were receive a two-dose schedule, 21 days apart, with 4 μg BBIBP-CorV inactivated SARS-CoV-2 vaccine. The primary safety outcome includes solicited local and systemic reactions prompted by and recorded in an electronic diary within 7 days post each injection, unsolicited adverse events and serious adverse events assessed from the receipt of each dose, and clinical laboratory abnormalities from dose 1 through 1month after dose 2. Laboratory tests included measurement of alanine aminotransferase, aspartate aminotransferase, serum total bilirubin, serum albumin, creatinine, blood urea nitrogen, and blood routine examination. Immunogenicity was assessed as the serum anti-SARS-CoV-2 specific antibody responses and neutralizing activity at 4 weeks after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations prior to any trial specific procedures.
* Male or female aged 18-59 years.

Exclusion Criteria:

* NA

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical workers in Ruijin Hospital who are willing to receive two dose of SARS-CoV-2 inactivated vaccine via intramuscular injection in the arm
Sampling Method: Probability Sample
Enrollment: 1370 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting local reactions | within 7days post each vaccination
  Pain at the injection site, swelling, itch, and redness
Percentage of participants reporting systemic events | within 7days post each vaccination
  Fever, headache, fatigue, nausea, vomiting, diarrhea, constipation, myalgia, arthralgia
Percentage of participants reporting adverse events | From Dose 1 through 1 month after Dose 2
  verified by investigators
Percentage of participants reporting serious adverse events | From Dose 1 through 1 month after Dose 2
  verified by investigators
Serum anti-SARS-CoV-2 speicfic antibody and neutralizing antibody titres | at 1 month after dose 2
  determination of anti-SARS-CoV-2 speicfic antibody and SARS-CoV-2 neutralizing antibody levels

SECONDARY OUTCOMES:
Serum anti-SARS-CoV-2 speicfic antibody and neutralizing antibody titres | at 6 months after dose 2
  determination of anti-SARS-CoV-2 speicfic antibody and SARS-CoV-2 neutralizing antibody levels
Serum anti-SARS-CoV-2 speicfic antibody and neutralizing antibody titres | at 12 months after dose 2
  determination of anti-SARS-CoV-2 speicfic antibody and SARS-CoV-2 neutralizing antibody levels

CONTACTS AND LOCATIONS:
Overall Officials: Erzhen Chen, Study Director — Ruijin Hospital; Xinxin Zhang, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital affiliated to Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu X, Wei D, Xu W, Liu C, Guo W, Li X, Tan W, Liu L, Zhang X, Qu J, Yang Z, Chen E. Neutralizing activity of BBIBP-CorV vaccine-elicited sera against Beta, Delta and other SARS-CoV-2 variants of concern. Nat Commun. 2022 Apr 4;13(1):1788. doi: 10.1038/s41467-022-29477-0. PMID 35379815